CLINICAL TRIAL: NCT00994786
Title: A Study of Pregabalin (Lyrica) Augmentation in Serotonin Reuptake Inhibitor-Refractory Obsessive Compulsive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Pfizer (Industry); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-273
Record Dates: First submitted 2009-10-05; First posted 2009-10-14 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: treatment-resistant; refractory; obsessive compulsive disorder; Lyrica; pregabalin; Serotonin Reuptake Inhibitor-Refractory Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pregabalin (Experimental)
  Interventions: Drug: pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pregabalin — pregabalin starting at 75 mg/day (at Study Week 0). Doses will be titrated up in 75 mg increments until a clinical response is achieved, as tolerated in the following manner: to 150 mg/day at the end of Study Week 1, to 225 mg/day at the end of Study Week 2, 300 mg/day at the end of Study Week 4, 450 mg/day at the end of Study Week 6 and to 600 mg/day at the end of Study Week 8. The maximum dose of pregabalin will be 600 mg/day.
  Other Names: Lyrica
  Arms: pregabalin
Drug: Placebo — Placebo starting at 75 mg/day (at Study Week 0). Doses will be titrated up in 75 mg increments until a clinical response is achieved, as tolerated in the following manner: to 150 mg/day at the end of Study Week 1, to 225 mg/day at the end of Study Week 2, 300 mg/day at the end of Study Week 4, 450 mg/day at the end of Study Week 6 and to 600 mg/day at the end of Study Week 8. The maximum dose of pregabalin/placebo will be 600 mg/day.
  Arms: Placebo

SUMMARY:
This study will examine the efficacy of pregabalin (Lyrica) added to SRI treatment in OCD for individuals who have not responded or only partially responded to an adequate trial of SRI. Although SRIs have demonstrated efficacy in OCD in numerous placebo-controlled trials, response rates have been as low as 40%. Augmentation strategies would be beneficial to maximize treatment response in OCD.

Pregabalin (Lyrica) is an anticonvulsant medication that appears to have a novel mechanism of action. It has been shown to enhance activity at gamma-amino-butyric acid (GABA) receptors as well as inhibit glutamate release. These two neurotransmitters systems have been implicated in the neurobiology of OCD.

The study will consist of patients who have not attained full response to an SRI. The patients will be randomized in a double-blind fashion to augmentation with pregabalin (Lyrica) or placebo. The dose of study medication will be flexible, starting at 75 mg/day and increasing in 75 mg increments to a maximum of 600 mg/day, based on efficacy and any side effects. Patients' response to treatment will be measured by the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS), the Montgomery Asberg Depression Rating Scale (MADRS), and the Clinical Global Impression Scale(CGI).

ELIGIBILITY:
Inclusion Criteria:

* Must be an outpatient with a primary DSM-IV Obsessive-Compulsive Disorder. Patients must have a score of greater than 20 on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS; Goodman et al., 1989b).
* Diagnosis of comorbid DSM-IV major depressive episode will be allowed in the study provided that the diagnosis is secondary to OCD, they have a baseline Montgomery Depression Rating Scale (MADRS) score of less than or equal to 19, and the onset of OCD predates the onset of the current episode of depression by five or more years.
* The ability to comprehend and comply with protocol requirements.
* Written consent must be provided prior to study entry.
* All women of childbearing potential (WOCBP) must be practicing a medically acceptable method of birth control
* All female subjects of childbearing potential (WOCBP), including those who are practicing a medically acceptable method of birth control, must have a negative serum pregnancy test within 72 hours prior to the start of study medication.

Exclusion Criteria:

* Patients with any other primary DSM-IV psychiatric diagnosis in addition to Obsessive Compulsive Disorder.
* Patients who currently fulfil criteria for DSM-IV eating disorder, body dysmorphic disorder, current alcohol or substance abuse, or who have a lifetime history of bipolar disorder. Patients with a history of Schizophrenia and other psychotic disorders, Delirium, Dementia, and Amnestic and other cognitive disorders.
* Subjects with a concurrent Axis II Cluster A Personality Disorder
* Borderline or Antisocial Personality Disorder.
* Subjects who based on history or mental status examination have a significant risk of committing suicide, in the investigator's opinion.
* Subjects with a history of more than three adequate trials with an SSRI.
* Subjects who have had an adequate trial of pregabalin.
* Subjects who have initiated psychotherapy in the last 4 months prior to the first visit.
* Subjects who, during the course of the study, would be likely to require treatment with prohibited concomitant therapy .
* Prior use of or a known allergy or hypersensitivity to pregabalin.
* Subjects who have participated in any clinical trial within 30 days prior to entering the study, or in a clinical trial involving a psychotropic medication within the 6 months prior to entering the study.
* Any subject who has been taking benzodiazepines before entering the study who: 1) cannot tolerate being free of benzodiazepines for 4 weeks, or 2) has signs or symptoms of benzodiazepine withdrawal or rebound at the end of those 4 weeks. Should a patient entering the study, who is currently on benzodiazepines develop discontinuation symptoms with discontinuation of their benzodiazepine, we will treat these symptoms with a more gradual benzodiazepine taper. Study will be delayed until the patient is able to tolerate the discontinuation for 4 weeks.
* Patients with a current seizure disorder, organic brain disorder or a history of seizure disorders (except for febrile seizures in childhood).
* Patients with thyroid pathology, the treatment of which has not been stabilized for at least three months.
* Patients on neuroleptic drugs in the two months prior to study entry or cognitive behavioural therapy specific to OCD within four weeks of study entry
* Pregnant or lactating females, or if sexually active and of childbearing potential, not using adequate methods of birth control.
* Patients with a history or evidence of a medical condition that would expose them to an increased risk of a significant adverse event or interfere with assessments of safety and efficacy during the trial.
* Patients receiving psychotropics of any kind, including betablockers and other anticonvulsants. Sleep medication such as oral chloral-hydrate or zopiclone are acceptable.
* Patients using any herbal psychoactive treatments, e.g. St John's Wort, Valerian, Kava Kava, L-tryptophan.
* Patients with any condition or on any therapy that, in the investigator's opinion, or as indicated in the pregabalin product label, may pose a risk to the subject.
* Patients who have had a major life event in the past three months, which in the judgement of the investigator is influencing their current condition.
* Patients having clinically significant abnormal laboratory, or ECG findings not resolved by further examinations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Yale-Brown-Obsessive-Compulsive-Scale | Baseline(Week 0) and Weeks 5, 9 and 12 (13 weeks)
Clinical Global Impression - Improvement | Weeks 1, 3, 5, 7, 9 and 12 (12 weeks)

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | Baseline (Week 0) (once - 1 week)
Sheehan Disability Scale | Baseline (Week 0) and Weeks 5, 9 and 12 (13 weeks)
Beck Depression Inventory | Weeks 1, 3, 5, 7, 9 and 12 (13 weeks)
Clinical Global Impression - Severity | Baseline (Week 0) and Weeks 1, 3, 5, 7, 9 and 12 (13 weeks)
Saving Inventory - Revised | Weeks 1, 5, 9 and 12 (12 weeks)
Dimensional Yale-Brown-Obsessive Compulsive Scale (D-Y-BOCS) | Baseline (Week 0) and Weeks 1, 5 and 12 (13 weeks)
Padua Inventory | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Van Ameringen, MD, FRCPC, Principal Investigator — McMaster Univeristy, Hamilton Health Sciences; Dan Stein, Principal Investigator — University of Stellenbosch
Locations (1):
- MacAnxiety Research Centre, Hamilton, Ontario, Canada

REFERENCES:
- See also: Related Info — http://www.macanxiety.com